CLINICAL TRIAL: NCT04414579
Title: The Efficacy and Safety of Faster Insulin Aspart (Fiasp®) Compared to Conventional Insulin Aspart (NovoLog®) as Correction Bolus in Patients With Type 1 Diabetes Using Continuous Subcutaneous Insulin Infusion (CSII) and Continuous Glucose Monitoring (CGM): a Cross-over Controlled Trial
Brief Title: The Efficacy and Safety of Faster Insulin Aspart (Fiasp®) Compared to Conventional Insulin Aspart (NovoLog®) as Correction Bolus
Acronym: PLATEAU
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mountain Diabetes and Endocrine Center (Other)
Responsible Party: Principal Investigator, Wendy Lane MD, Wendy Lane, MD, Principal Investigator, Mountain Diabetes and Endocrine Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GPP2019
Record Dates: First submitted 2020-05-26; First posted 2020-06-04 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: continuous glucose monitoring; continuous subcutaneous insulin infusion; hyperglycemia; correction bolus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hyperglycemia | interventions — Insulin Aspart

STUDY DESIGN:
Intervention Model Description: This is a 25-week open-label prospective single center 2 arm crossover trial consisting of a CSII settings (basal, bolus, and correction factors) will be optimized for a 2-week run in period followed by a 10-week period of CSII use with the assigned insulin. After a 12-week maintenance period, each group will cross over to the other insulin (conventional insulin aspart or Fiasp) by CSII for a second 2-week optimization period followed by a 10-week treatment period.
Masking Description: This is an open-label crossover trial. Subjects will be randomized to treatment sequence (Fiasp then NovoLog or NovoLog then Fiasp), each for a 12-week treatment period, by CSII. Randomization sequence will be determined by computerized randomization program. All patients will receive both treatments unless they drop out. Dropouts are unlikely since the participants are all regular continuing patients of the site's clinical practice.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- No Intervention: Conventional Insulin Aspart (NovoLog®) (No Intervention): In the aspart group, the subject will only take aspart through the their pump. This study population will have an established expertise in diabetes self-management with previous knowledge of insulin pump therapy and Dexcom Continuous Glucose Monitoring (CGM). Allowing the subjects to use their insulin pumps for bolus insulin delivery, as they are accustomed, will minimize the chances of skipping meal boluses and correction doses. Aspart is put into their pump and delivered to their body through a small tube placed under your skin. In this NovoLog®-only treatment group, the subject will take aspart with each meal while your pump also gives you a slow, continuous dose of aspart for basal insulin. This treatment group is very similar (or even identical) to the treatment the subject was receiving prior to starting the study.
- Faster Insulin Aspart (Fiasp®) (Active Comparator): In the Fiasp group, the subject will only take aspart through the their pump. This study population will have an established expertise in diabetes self-management with previous knowledge of insulin pump therapy and Dexcom Continuous Glucose Monitoring (CGM). Allowing the subjects to use their insulin pumps for bolus insulin delivery, as they are accustomed, will minimize the chances of skipping meal boluses and correction doses. Fiasp is put into their pump and delivered to their body through a small tube placed under their skin. In this Fiasp treatment group, the subject will take fiasp with each meal while their pump also gives them a slow, continuous dose of aspart for basal insulin. This treatment group is very similar (or even identical) to the treatment the subject was receiving prior to starting the study.
  Interventions: Drug: Faster Insulin Aspart (Fiasp®)

INTERVENTIONS:
Drug: Faster Insulin Aspart (Fiasp®) — Subjects will be randomized either to use Fiasp or conventional insulin aspart in CSII. CSII settings (basal, bolus, and correction factors) will be optimized using a meal challenge for a 2-week run in period followed by a 10-week period of CSII use with the assigned insulin. After a 12-week maintenance period, each group will cross over to the other insulin (conventional insulin aspart or Fiasp) by CSII for a second 2-week optimization period followed by a 10-week treatment period.
  Other Names: Conventional Insulin Aspart (NovoLog®)
  Arms: Faster Insulin Aspart (Fiasp®)

SUMMARY:
The purpose of this investigator-initiated trial is to compare the efficacy in terms of time to recovery from hyperglycemia as measured by time to arrest of hyperglycemic excursion ("glucose plateau point", primary endpoint) and return to premeal glucose target if feasible (secondary endpoint) between Fiasp and conventional insulin aspart when used as a correction bolus. These endpoints will be determined by CGM (Dexcom) from data exported from the Dexcom Clarity program.

DETAILED DESCRIPTION:
Patients with type 1 DM using CSII require bolus insulin for two purposes: first, to cover carbohydrate intake to control postprandial glucose, and second, to correct episodes of hyperglycemia. The latter function is referred to as a "correction dose" or "correction bolus". Insulin pumps have bolus calculators which calculate correction doses based on the patient's individualized BG target and insulin sensitivity factor (ISF). Rapid-acting insulin analogues delivered by pump typically require 2 to 4 hours to fully correct an acute hyperglycemic episode, and sometimes multiple correction doses are needed to normalize the blood glucose level. This can be frustrating for patients, particularly when a correction bolus is necessary in addition to a meal bolus; frequently, patients must wait for the correction bolus to take effect and delay eating until the blood glucose has begun to normalize to avoid severe postprandial hyperglycemia. There is consequently an unmet need in insulin delivery, and in particular in CSII, for an insulin which can correct a hyperglycemic episode more rapidly than is currently possible with rapid-acting insulin analogues.

Faster insulin aspart (Fiasp) is a novel formulation of insulin aspart with an accelerated time-action profile which results in twice the exposure to insulin and 74% greater insulin action within the first 30 minutes after injection compared to conventional insulin aspart. This results in twice-as-fast onset of appearance in the bloodstream (4 vs. 9 min compared to conventional insulin aspart) which has been demonstrated to reduce postprandial glucose levels in patients with type 1 DM using CSII. Theoretically, this faster insulin action would be useful in correction dosing during acute episodes of hyperglycemia to normalize the blood glucose level more rapidly than is currently possible with conventional insulin aspart (NovoLog).

Many patients with type 1 DM using CSII now also use continuous glucose monitoring (CGM) for making insulin dosing decisions. Currently the FDA has approved 2 CGM systems for nonadjunctive use in bolus insulin dose calculations. Only one of these systems, the Dexcom, reads continuously to the patient and has alarms to warn of impending episodes of hyper- or hypoglycemia, and this is the system used most commonly by patients with type 1 DM using open-loop CSII. Patients now incorporate the Dexcom trend arrow, which depicts the rate and direction of glucose change, into the correction dose calculation, and recommendations on how to incorporate CGM information into correction dose calculations have recently been updated based on an expert consensus report. However, these guidelines were created for use with rapid acting insulin analogues. How they might need to be modified for use with Fiasp (the first and only ultra-rapid insulin analogue) is not known.

The purpose of this investigator-initiated trial is to compare the efficacy in terms of time to recovery from hyperglycemia as measured by time to arrest of hyperglycemic excursion ("glucose plateau point", primary endpoint) and return to premeal glucose target if feasible (secondary endpoint) between Fiasp and conventional insulin aspart when used as a correction bolus. These endpoints will be determined by CGM (Dexcom) from data exported from the Dexcom Clarity program.

Study hypothesis:

Compared to conventional insulin aspart, Fiasp will correct hyperglycemia (defined as arrest of rise of blood glucose, following correction bolus, ie, GPP ) faster than conventional insulin aspart in subjects with type 1 DM using CSII.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients > 18 years of age
* Type 1 DM of > 1 year duration
* Use of any open loop insulin pump, Tandem T-Slim with Basal IQ, Insulet Omnipod Dash, or any other investigator-approved insulin pumps with Dexcom CGM G5, G6, or newer version for > 6 months
* Good baseline glycemic control (HbA1c < 7.5%; low risk of hypoglycemia by CGM as defined by Dexcom Clarity report)
* No episodes of severe hypoglycemia in the previous 3 months
* Pump download shows regular meal bolusing, accurate carbohydrate counting ability, and willingness to use exercise markers in Dexcom
* CGM download shows regular use (>85% of time) and regular calibration if using G5 sensor (G6 requires no calibration)
* Females using adequate contraception

Exclusion Criteria:

* Use of CGM other than Dexcom G5 or G6 or a newer Dexcom CGM version
* Suboptimal baseline glycemic control (HbA1c > 7.5%)
* Pump or CGM download shows suboptimal use of devices (lack of meal boluses, frequent overrides of pump, excessive pump suspension, inadequate calibration or inconsistent usage of CGM)
* Serious comorbidities including CVD with recent event, actively treated malignancy, renal dysfunction with eGFR < 45 ml/min, or any other condition which in the opinion of the investigator would preclude subject's ability to participate in trial
* Females unwilling to use contraception, planning pregnancy or breastfeeding
* Use of any other glucose-lowering agents than insulin
* Hypersensitivity to insulin aspart or one of the excipients in faster insulin aspart
* Known diabetic gastroparesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-03-27 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Time to stabilization of rising blood sugar by CGM after correction bolus | 2 weeks
  Time (in minutes) to stabilization of rising blood sugar (GPP) by CGM after correction bolus during the final 2 week maintenance period. Two categories of correction dose will be analyzed: 1) those following an isolated correction dose (taken independently of a meal dose), and 2) those taken as part of a combination bolus with a meal dose.

SECONDARY OUTCOMES:
Incidence of early hypoglycemia | 25 weeks
  Incidence of early hypoglycemia (Blood glucose < 54 mg/dl within 1 and 2 hours) following correction bolus with each insulin (Key Safety Endpoint)
Change in Insulin Sensitivity Factor | 25 weeks
  Change in Insulin Sensitivity Factor, if any, required for hypoglycemia prevention using Fiasp as recorded by continuous subcutaneous insulin infusion device setting report
Change in Insulin On Board | 25 weeks
  Change in Insulin On Board, if any, required for prevention of late hyperglycemia using Fiasp as recorded by continuous subcutaneous insulin infusion device setting report
GlycoMark differences between arms | 25 weeks
  GlycoMark (1,5 anhydroglucitol, a marker of postprandial glucose excursion) during use of each insulin.
HbA1c differences between arms | 25 weeks
  HbA1c during use of each insulin
Percent time spent in target range, hyperglycemic range, and hypoglycemic range | 4 weeks
  Percent time spent in target range, hyperglycemic range and hypoglycemic range by Continuous Glucose Monitoring (CGM) on each insulin during the final 2 weeks of each treatment period. Target ranges include 70-180 mg/dL. Hyperglycemia ranges to be captured will include Category 1: 181-250 mg/dL and Category 2: above 250 mg/dL. Hypoglycemia ranges to be captured include Category 1: 69-54 mg/dL and Category 2: below 54 mg/dL.
Standard deviation differences between arms | 4 weeks
  Standard deviation of mean blood glucose as determined by CGM on each insulin
Treatment related impact measures between arms | 6 weeks
  Treatment related impact measures on each insulin using TRIM D questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Mountain Diabetes and Endocrine Center, Asheville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and statistical analysis will be available to any researcher with appropriate request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: post-study, up to 5 years
Access Criteria: email Principal Investigator

REFERENCES:
- [Background] Bode BW, Johnson JA, Hyveled L, Tamer SC, Demissie M. Improved Postprandial Glycemic Control with Faster-Acting Insulin Aspart in Patients with Type 1 Diabetes Using Continuous Subcutaneous Insulin Infusion. Diabetes Technol Ther. 2017 Jan;19(1):25-33. doi: 10.1089/dia.2016.0350. Epub 2017 Jan 5. PMID 28055230
- [Background] Aleppo G, Laffel LM, Ahmann AJ, Hirsch IB, Kruger DF, Peters A, Weinstock RS, Harris DR. A Practical Approach to Using Trend Arrows on the Dexcom G5 CGM System for the Management of Adults With Diabetes. J Endocr Soc. 2017 Nov 20;1(12):1445-1460. doi: 10.1210/js.2017-00388. eCollection 2017 Dec 1. PMID 29344577
- [Background] Heise T, Pieber TR, Danne T, Erichsen L, Haahr H. A Pooled Analysis of Clinical Pharmacology Trials Investigating the Pharmacokinetic and Pharmacodynamic Characteristics of Fast-Acting Insulin Aspart in Adults with Type 1 Diabetes. Clin Pharmacokinet. 2017 May;56(5):551-559. doi: 10.1007/s40262-017-0514-8. PMID 28205039
- [Background] Russell-Jones D, Bode BW, De Block C, Franek E, Heller SR, Mathieu C, Philis-Tsimikas A, Rose L, Woo VC, Osterskov AB, Graungaard T, Bergenstal RM. Fast-Acting Insulin Aspart Improves Glycemic Control in Basal-Bolus Treatment for Type 1 Diabetes: Results of a 26-Week Multicenter, Active-Controlled, Treat-to-Target, Randomized, Parallel-Group Trial (onset 1). Diabetes Care. 2017 Jul;40(7):943-950. doi: 10.2337/dc16-1771. Epub 2017 Mar 29. PMID 28356319
- [Background] Bergenstal RM, Garg S, Weinzimer SA, Buckingham BA, Bode BW, Tamborlane WV, Kaufman FR. Safety of a Hybrid Closed-Loop Insulin Delivery System in Patients With Type 1 Diabetes. JAMA. 2016 Oct 4;316(13):1407-1408. doi: 10.1001/jama.2016.11708. No abstract available. PMID 27629148
- [Background] Klonoff DC, Evans ML, Lane W, Kempe HP, Renard E, DeVries JH, Graungaard T, Hyseni A, Gondolf T, Battelino T. A randomized, multicentre trial evaluating the efficacy and safety of fast-acting insulin aspart in continuous subcutaneous insulin infusion in adults with type 1 diabetes (onset 5). Diabetes Obes Metab. 2019 Apr;21(4):961-967. doi: 10.1111/dom.13610. Epub 2019 Jan 13. PMID 30537180

DOCUMENTS (1):
  • Study Protocol (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/79/NCT04414579/Prot_000.pdf